CLINICAL TRIAL: NCT01357421
Title: A Phase 1 Double-blind, Randomized, Placebo-controlled Study Evaluating the Effects of a Single Intravenous Dose of TT301 on LPS-induced Changes in Blood Cytokine Levels in Healthy Male Volunteers
Brief Title: Effects of TT301 on Cytokine Levels Post Endotoxin Challenge
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMX-103
Record Dates: First submitted 2011-05-13; First posted 2011-05-20 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TT301 (Experimental): Investigational drug TT301
  Interventions: Drug: TT301
- Placebo (Placebo Comparator): Normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TT301 — Single iv dose of TT301
  Other Names: TT301 iv
  Arms: TT301
Drug: Placebo — Single iv dose of 0.9% sodium chloride for injection USP
  Other Names: 0.9% sodium chloride for injection USP
  Arms: Placebo

SUMMARY:
This study will evaluate the effects of TT301 on cytokine levels in healthy male volunteers participating in an endotoxin challenge.

DETAILED DESCRIPTION:
The LPS human endotoxemia model results in a well characterized, transient acute inflammatory response. The model has been widely used for decades as a system to study new therapeutic agents for inflammation before wider clinical studies are undertaken. This study will evaluate the effects of TT301 on cytokine levels in healthy male volunteers participating in an endotoxin challenge.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18 to 40 years, inclusive
* 55 - 95 kg, inclusive

Exclusion Criteria:

* Evidence of any clinically significant disease
* History of cancer
* History of syncope or severe vasovagal events
* Antibiotic treatment within 60 days of Day 1
* Surgical procedure within 60 days of Day 1
* Hepatitis C, Hepatitis B
* Tuberculosis
* HIV
* Requirement for medications (prescription/OTC) during the study
* Donated > 250 mL blood within 30 days of Day 1
* Donated > 750 mL blood within 60 days of Day 1
* In a clinical trial of an immunosuppressive drug within 6 months of Day 1
* Received any vaccination within 6 months of Day 1
* Any clinically important allergy
* Known allergy/sensitivity to lactose and/or polyethylene glycol

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Cytokine levels post LPS challenge | Measured up to 12h post-LPS

CONTACTS AND LOCATIONS:
Overall Officials: Laura Agensky, BSc, MBA, Study Director — Transition Therapeutics Inc. / Waratah Pharmaceuticals Inc.
Locations (1):
- Duke Clinical Research Unit, Durham, North Carolina, United States